CLINICAL TRIAL: NCT06532422
Title: Study of Post-operative Complications After Laparoscopic Outpatient Nephrectomy in Patients With Localised Kidney Cancer
Brief Title: Study of Post-operative Complications After Laparoscopic Outpatient Nephrectomy
Acronym: NEPHRAMBU
Status: Recruiting | Type: Observational
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023-A02569-36
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cohort of outpatients: Adult patients diagnosed with localised kidney cancer, undergoing scheduled surgery for partial or total laparoscopic nephrectomy on an outpatient basis.
  Interventions: Procedure: Partial or total laparoscopic nephrectomy

INTERVENTIONS:
Procedure: Partial or total laparoscopic nephrectomy — Nephrectomy is currently the primary indication for localised kidney cancer. All patients consulting a surgeon at the Clinique de la Sauvegarde for localised kidney cancer, for which surgical excision has been validated by the multidisciplinary consultation meeting and who are eligible for outpatient treatment, will be offered the opportunity to take part in this study during the preoperative consultation.

SUMMARY:
The purpose of this study is to compare to assess the incidence of post-operative complications related to nephrectomy, which occur up to 1 month after the operation.

DETAILED DESCRIPTION:
This is an observational, prospective, open, non-comparative (single arm), single-centre study.

The study population consisted of adult patients diagnosed with localised kidney cancer and scheduled for outpatient partial or total laparoscopic nephrectomy.

Patients eligible for outpatient surgery will be identified during the initial consultation with the urological surgeon. When the indication for surgery has been validated at the multidisciplinary consultation meeting and is planned to be performed as an outpatient procedure, the study will be proposed to the patient by the investigator during the preoperative consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 ;
* Localised kidney cancer ;
* Validation of curative treatment at a multidisciplinary consultation meeting;
* Partial or total laparoscopic nephrectomy scheduled on an outpatient basis;
* Membership of a social security scheme or receiving State Medical Aid;
* Patient able to understand the information relating to the study, to read the information leaflet and who has given his/her oral non-objection.

Exclusion Criteria:

* Emergency intervention ;
* Patient not eligible for outpatient treatment;
* Long-term curative anti-coagulant treatment ;
* Resident more than 100km from the clinic;
* Home alone on the first night;
* Patient of protected age (under guardianship or curatorship, or deprived of liberty).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with localised kidney cancer, undergoing scheduled surgery for partial or total laparoscopic nephrectomy on an outpatient basis.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-12-13 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of complications | 1 month
  The study will observe the incidence and describe the type, number, severity, duration and frequency of complications that may arise in the immediate post-operative period following ambulatory nephrectomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique de la Sauvegarde, Lyon, France